CLINICAL TRIAL: NCT00898261
Title: Genetic Risk Classes in Adult Acute Lymphocytic Leukemia
Brief Title: Gene Expression in Tissue From Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000526268; ECOG-E2993T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia | interventions — Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: flow cytometry

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at gene expression in tissue from patients with acute lymphoblastic leukemia enrolled in clinical trial ECOG-2993.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify genes involved in specific biologic processes or molecular functions that contribute to the mechanisms by which the BCR/ABL tyrosine kinase induces a leukemic phenotype using RNA banked from patients with BCR/ABL-positive acute lymphoblastic leukemia (ALL) enrolled on ECOG-2993.
* Compare patterns of mRNA expression of BCR/ABL fusion protein in patients with B-lineage ALL vs patients with ALL and no cytogenetic abnormalities enrolled on ECOG-2993.
* Determine both shared and differing expression patterns in patients with BCR/ABL-positive and cytogenetically negative ALL with respect to achievement of complete remission and duration of disease-free and overall survival.

OUTLINE: This is a multicenter study.

Total RNA is isolated from stored tissue samples and integrity is verified by reverse transcription-polymerase chain reaction (RT-PCR). cDNA libraries are created from total RNA and gene expression is analyzed via microarray analysis.

Genes of interest are further analyzed by flow cytometry and RT-PCR.

PROJECTED ACCRUAL: A total of 137 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of acute lymphoblastic leukemia
* Tissue banked on protocol ECOG-2993 meeting the following criteria:

  * Leukemic blast cell population immunophenotyped in detail (e.g., including CD25) in ECOG's Immunophenotyping Reference Laboratory
  * Flow cytometric analysis of gated blast cells reveals association with the B-cell lineage
  * Mononuclear cell fraction used for RNA isolation contains 75-99% blasts (median 85%)
  * Negative for TEL/AML1, MLL/AF4, and E2A/PBX1 by qualitative reverse transcription-polymerase chain reaction (RT-PCR)
  * No FLT3 gene mutations
  * BCR/ABL-positive samples meeting the following criteria:

    * Presence of t(9;22)(q34;q11) by standard cytogenetics
    * Detection of either p190 BCR/ABL or p210 BCR/ABL transcripts by qualitative RT-PCR
  * Patients with genetic risk factors must meet the following criterion:

    * Only a normal diploid karyotype is present in ≥ 15 metaphases by standard cytogenetics

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E2993
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2007-10-26 (Actual); Primary Completion 2012-07-19 (Actual); Study Completion 2012-07-19 (Actual)

PRIMARY OUTCOMES:
Genes involved in specific biologic processes or molecular functions that contribute to the mechanisms by which the BCR/ABL tyrosine kinase induces a leukemic phenotype | 1 month
Comparison of patterns of mRNA expression of BCR/ABL fusion protein in patients with B-lineage acute lymphoblastic leukemia (ALL) vs patients with ALL who lack cytogenetic abnormalities | 1 month
Shared and differing expression patterns in patients with BCR/ABL-positive and cytogenetically negative ALL with respect to achievement of complete remission and duration of disease-free and overall survival | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Paietta, PhD, Study Chair — Our Lady of Mercy Medical Center